CLINICAL TRIAL: NCT05392426
Title: High-sensitive Troponin I Increase After Surgery is Associated With Left Ventricular Global Longitudinal Strain Among Patients With Elderly Coronary Heart Disease
Brief Title: Left Ventricular Global Longitudinal Strain and Postoperative Myocardial Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: GLS and Myocardial injury
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood will be collected for biochemical testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Left Ventricular Global Longitudinal Strain — Left Ventricular Global Longitudinal Strain is collected from Speckle tracking imaging (STI) technique of echocardiography. This index is tested before and after the surgery.
Device: EF CO SV EDV ESV — Ejection fraction、cardiac output、stroke volume、end diastolic volume、end systolic volume. These indexes are collected before and after the surgery, using traditional echocardiography.

SUMMARY:
To use left ventricular global longitudinal strain as a means of monitoring myocardial exercise function during anaesthesia in patients with coronary artery disease, to explore the association with the occurrence of postoperative myocardial injury, and to perform a predictive study of postoperative myocardial injury. The study was designed according to a prospective follow-up cohort.

DETAILED DESCRIPTION:
The incidence and risk of postoperative myocardial injury in patients with coronary artery disease is high, and there is no definitive monitoring tool to predict postoperative myocardial injury. Speckle tracking imaging (STI), which quantifies strain and ventricular torsion in all segments of the heart, is more sensitive to subtle changes in myocardial contractility than conventional ultrasound. This project proposes to use 4D-STI as a means of monitoring myocardial exercise function during anaesthesia in patients with coronary artery disease, to explore the association with the occurrence of postoperative myocardial injury, and to perform a predictive study of postoperative myocardial injury. The study was designed according to a prospective follow-up cohort. The protocol was developed with reference to the STROBE guidelines for cohort studies. In this study, 2.5 ml of venous blood specimens were collected before surgery and at the end of surgery and sent to the laboratory. Intraoperative data collection was performed in the operating theatre and follow-up was obtained on the ward and during telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-90;
2. According to the European Heart Association's diagnostic criteria for chronic coronary syndrome in 2019.Patients with suspected coronary heart disease and stable angina pectoris, with or without dyspnea; New heart failure or left ventricular dysfunction, suspected coronary heart disease; Patients with acute coronary syndrome who are asymptomatic or stable within one year of onset, or who will undergo revascularization in the near future;Patients with an initial diagnosis or revascularization for more than one year, with or without symptoms; Angina pectoris, suspected vasospasm, or microvascular disease patients; During screening, asymptomatic people with coronary heart disease were discovered;
3. ASA II~III; NYHA II~III; require general anesthesia;
4. no history of anesthetic allergy;
5. agreed to participate in the study and signed the informed consent form.

Exclusion Criteria:

1. Congenital heart disease, severe ventricular arrhythmia, atrial fibrillation, severe valvular regurgitation;
2. Severe history of chronic obstructive pulmonary illness (COPD severity III or IV), individuals with severe or uncontrolled bronchial asthma, pulmonary infection, bronchiectasis;
3. Patients with persistent drinking and known or suspected abusers of other narcotic analgesics;
4. Obese (BMI 30 kg/m2)
5. Cardiac surgical procedures are planned.

Ages: 65 Years to 90 Years | Sex: All
Age Groups: Older Adult
Study Population: According to the European Heart Association's diagnostic criteria for chronic coronary syndrome in 2019, refers to the many stages of coronary heart disease other than the clinical manifestations dominated by acute coronary thrombosis.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative high-sensitive troponin I change | 15 minutes after the ending of the surgery
  high-sensitive troponin I will be tested before and after surgery

SECONDARY OUTCOMES:
Incidence of postoperative arrhythmia events | from the ending of surgery to 72 hours after surgery
  postoperative arrhythmia events are recorded according to follow-up visits after surgery
Incidence of postoperative myocardial infarct events | from the ending of surgery to 72 hours after surgery
  postoperative myocardial infarct events are recorded according to follow-up visits after surgery

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — The Second Affiliated Hospital, Chongqing Medical University
Locations (2):
- China (2):
  - Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality
  - The second affiliated hospital of Chongqing medical university, Chongqing

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within five years